CLINICAL TRIAL: NCT03377829
Title: A Multicenter Prospective Controlled Trial of Laser Ablation Versus Surgery for the Treatment of Papillary Thyroid Microcarcinoma
Brief Title: A Multicenter Trial of PLA vs. Surgery for Treating PTMC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: WeiWei Zhan (Other)
Responsible Party: Sponsor-Investigator, WeiWei Zhan, Director, Head of Ultrasound Department; Clinical Professor, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1001253709008902933
Record Dates: First submitted 2017-11-26; First posted 2017-12-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Thyroid Cancer; Treatment Related Cancer
Keywords: Papillary Thyroid Microcarcinoma; Percutaneous Laser Ablation; thyroidectomy; ultrasonography; double-blind
MeSH Terms: conditions — Thyroid Neoplasms; Neoplasms, Second Primary; Papillary Thyroid Microcarcinoma

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous laser ablation(PLA) (Experimental): Eligible participants with PTMC will be randomly assigned to this group and undergo percutaneous laser ablation(PLA). All the process is under the detection of real-time ultrasound.After surgery, all the patients will accept contrast-enhanced ultrasound(CEUS), regular ultrasound follow-up, thyroid functional detection, fine-needle aspiration biopsy(FNAB), neck CT.Per and post-operative complications, need of drug treatment, length of hospital admission and customer satisfaction will be registered.
  Interventions: Procedure: PLA
- Surgery (Active Comparator): Eligible participants with PTMC will be randomly assigned to this group and undergo total/subtotal thyroid surgery.
  Interventions: Procedure: Thyroid Surgery

INTERVENTIONS:
Procedure: PLA — During the PLA, the patient is in supine position with head extended: the physician, ultrasound assistant and trained nurse work within the sterile field. Under constant ultrasound image guidance and after local anesthesia by means of 2% xylocaine infiltration, thin needles (21G) are positioned in the thyroid lesion, within safety distance from the surrounding anatomical structures. A plane-cut tip fiber optics is inserted into the PTMC through the needle. The laser at 1064 nm wavelength is turned on for 10 minutes until the pre-established energy dose is attained. There is usually no pain or very limited pain.
  Arms: Percutaneous laser ablation(PLA)
Procedure: Thyroid Surgery — Patients are routinely disinfected and spread the drapes after general anesthesia. Neck skin, fat, placenta muscle are incised successively. The flap is separated to the upper edge of thyroid cartilage, neck white line is incised and anterior muscle group is separated. Then both sides thyroid lobes are exposed. Cut off the isthmus, ligature the thyroid artery, cut off the upper pole. Ligature and cut off the ipsilateral thyroid vein. Reveal and protect the ipsilateral recurrent laryngeal nerve and the parathyroid gland during the entire process. Finally patient is performed total thyroidectomy or subtotal thyroidectomy.
  Arms: Surgery

SUMMARY:
This is a multicenter prospective controlled trial of percutaneous laser ablation(PLA) versus conventional surgery for the treatment of papillary thyroid microcarcinoma (PTMC).

DETAILED DESCRIPTION:
PLA is the acronym for "Percutaneous Laser Ablation". The treatment consists in the destruction (ablation) of Papillary Thyroid Micro Carcinoma by means of optical fibers that deliver high-energy light (laser) into the lesion through skin puncturing (percutaneous). The procedure is performed under ultrasound imaging guidance (ultrasound-guided). The destruction of the lesion occurs through overheating and coagulation. PLA, however, still needs a large-scale validation trial in order to be considered as an effective alternative to both surgery or follow-up for low-risk PTMC in elderly patients and/or in patients with co-morbidities that might expose the patients to a high surgical risk.

After a comprehensive information, patients will be consecutively assigned to Group 1 (surgery, preferentially lobectomy) or to Group 2 (percutaneous laser ablation, performed according to the attached procedure).Peri and post-operative complications, need of drug treatment, length of hospital admission and customer satisfaction will be registered.

The aims of this study are as follows: 1.To establish the rate of cure or partial ablation; 2.To compare the complication rate, time expenditure and costs of two procedures; 3.To assess changes in thyroid function and the need of substitution therapy with two procedures; 4.To assess the tolerability of the procedure, the customer satisfaction and the impact on the quality of life of the patients between conventional surgery and PLA.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed PTMC (maximun diameter> = 5 mm and < = 10 mm) proved by fine needle aspiration biopsy with good thyroid function;
* Age≥ 18 Y;
* Single nodule without thyroid capsule contact;
* There had more than 3mm distance between nodules and trachea, carotid artery, recurrent laryngeal nerve (The distance should up to 5mm after injection of isolation fluid);
* No coarse calcification or eggshell-like calcification;
* Imaging examination without local or distant metastasis;
* Without chemotherapy, radiotherapy and other related therapies;
* A complete clinical, pathological and follow-up information;
* Get informed consent signed by the patient or family member.

Exclusion Criteria:

* Multifocal PTMC;
* Combined with other types of thyroid cancer or hyperthyroidism;
* Lesion contact with thyroid capsule or located in the isthmus;
* Serious coagulation dysfunction;
* Contralateral vocal cord paralysis;
* Imaging examination with local or distant metastasis;
* Active Tuberculosis and HIV-positive patients;
* Patients can not understand or follow research protocol;
* Pregnant woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Serological examination of thyroid function | up to 12 months
  Hyperthyreosis or hypothyroidism.

SECONDARY OUTCOMES:
Recurrence rate | up to 12 months
  The recurrence rate in the thyroid bed or regional lymph-nodes
Therapeutic Effect | up to 24 months
  The rate of cure (defined as the absence of disease persistence at US examination and FNAB) between two methods.

CONTACTS AND LOCATIONS:
Overall Officials: WeiWei Zhan, Ph.D, Principal Investigator — Ruijin Hospital, affiliated to Medical School of Shanghai Jiaotong University
Locations (13):
- China (11):
  - Ultrasound Department, Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Ultrasound Department of the Third Hospital Affiliated to Zhongshan University, Guangzhou, Guangdong
  - Ultrasound Department, the Second Affiliated Hospital of Harbin Medical Univercity, Harbin, Heilongjiang
  - Ultrasound Department, the Xiangya Third Hospital of Zhongnan University, Changsha, Hunan
  - Ultrasound Department, the First Affliction Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Ultrasound Department, the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Ultrasound Department, First people's Hospital Affiliated to Medical School of Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Ultrasound Department, Ruijin Hospital Affiliated to Medical School of Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - The department of ultrasound ,second affiliated hospital of xi'an jiaotong university, Xi’an, Shanxi
  - Department of Ultrasonography, Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Department of Ultrasound Medicine, the First Hospital Affiliated to Medical School of Zhejiang University, Hangzhou, Zhejiang
- Italy (2):
  - Department of Endocrinology, Regina Apostolorum Hospital, Rome
  - Diagnostic Imaging, Regina Apostolorum Hospital, Rome